CLINICAL TRIAL: NCT06707298
Title: The Role of Multidetector Computed Tomography(MDCT) in Grading of Oesophageal Varices in Cirrhotic Patients in Comparison to Endoscopy
Brief Title: Role of MDCT in Grading of Esophageal Varices
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Saad Wally, Resident Doctor, Assiut University
Other Study IDs: MDCT in esophageal varices
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: MDCT Esoghageal Varices
Keywords: MDCT; Esophageal varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Esophageal varices are one of the major complications of liver cirrhosis.Accurate grading of these varices is essential for effective management . Traditionally, esophagogastroduodenoscopy is the gold standard for diagnosing and grading esophageal varices,Multi detector computed tomography (MDCT) has emerged as a non-invasive alternative for evaluating esophageal varices.it particularly appealing for patients who contraindicated to endoscopy .

DETAILED DESCRIPTION:
Esophageal varices are one of the major complications of liver cirrhosis, with an estimated prevalence of approximately 80% with decompensated patients and 50% in compensated cirrhosis, pose a significant risk of life-threatening of bleeding due to portal hypertension. Accurate grading of these varices is essential for effective management . Traditionally, esophagogastroduodenoscopy (EGD) is the gold standard for diagnosing and grading esophageal varices . IT provides direct visualization, allowing for detailed assessment of variceal size and other risk factors for bleeding . However, it is an invasive procedure that requires sedation and carries some risks, such as bleeding or perforation .

Multi detector computed tomography (MDCT) has emerged as a non-invasive alternative for evaluating esophageal varices. It offers detailed cross-sectional images and is widely available, providing a broader assessment of abdominal pathology. Its non-invasive nature makes it particularly appealing for patients who contraindicated to endoscopy .

ELIGIBILITY:
Inclusion Criteria:

-Cirrhotic patients with portal hypertension undergoing upper GI endoscopy.

Exclusion Criteria:

-Contraindication to contrast:( severe renal insufficiency, allergy to contrast agents).

-Previous history of upper GI endoscopy with intervention (band ligation or sclerotherapy).-

* Pregnancy.
* Patients with previous transjagular intrahepatic portosystemic shunt (TIPS).
* Patients with contraindication to endoscopy (severe cardiopulmonary conditions, coma "unless the patient is intubated", and cardiac arrhythmias)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic pateints with esophageal varices with no previous history of intervention andnot contraindicated to endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between CT and endscopy in esophageal varices | Baseline
  Agreement between MDCT and endoscopy in the grading of esophageal varices

SECONDARY OUTCOMES:
Assessment other complication of varicesand cirrhosis in CT | Baseline
  Assessment of the presence of complications or additional findings (e.g., portal vein thrombosis,Liver pathology) and other complication related to portal hypertension as ascites or splenomegaly on MDCT.

REFERENCES:
- [Background] Kumar R, Nandolia KK, Sharma P, Bhadoria AS, Chauhan U, Patnaik I, Saxena S. Computed tomography virtual oesophagography for the grading of oesophageal varices in cirrhotic liver disease patients with upper gastrointestinal endoscopic examination as the gold standard: a diagnostic validation study. Pol J Radiol. 2023 Apr 5;88:e187-e193. doi: 10.5114/pjr.2023.126459. eCollection 2023. PMID 37234460
- [Background] Li J, Zhu Y, Ni J, Wang L, Lei J. Computed tomography for the diagnosis of gastroesophageal varices and risk assessment in patients with cirrhosis: a systematic review and meta-analysis. Diagn Interv Radiol. 2024 Nov 6;30(6):335-350. doi: 10.4274/dir.2024.242723. Epub 2024 May 20. PMID 38767277
- [Background] Zhang YH, Hu B. Future directions of noninvasive prediction of esophageal variceal bleeding: No worry about the present computed tomography inefficiency. World J Gastrointest Endosc. 2024 Mar 16;16(3):108-111. doi: 10.4253/wjge.v16.i3.108. PMID 38577650
- [Background] Gunda DW, Kilonzo SB, Mamballah Z, Manyiri PM, Majinge DC, Jaka H, Kidenya BR, Mazigo HD. The magnitude and correlates of esophageal Varices among newly diagnosed cirrhotic patients undergoing screening fibre optic endoscope before incident bleeding in North-Western Tanzania; a cross-sectional study. BMC Gastroenterol. 2019 Nov 29;19(1):203. doi: 10.1186/s12876-019-1123-9. PMID 31783802